CLINICAL TRIAL: NCT05705037
Title: Molar Incisor Hypomineralization and Hypersensitivity in Paediatric Age: a Comparison of Treatment Protocols
Brief Title: MIH and Hypersensitivity in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Elena Bardellini, Associated Professor, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIH-2020.1
Record Dates: First submitted 2023-01-21; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Dentin Sensitivity; Molar Incisor Hypomineralization
Keywords: Photobiomodulation; CPP-ACPF; Dentin; Hypersensitivity; Children
MeSH Terms: conditions — Dentin Sensitivity; Molar Hypomineralization; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (CPP-ACPF mousse + sham light therapy) (Sham Comparator): CPP-ACPF mousse (MI Paste®) was applied with a microbrush on the cervical buccal surface of each tooth for 5 minutes and it was subsequently distributed for 20 seconds with a rubber cup coupled to a low speed handpiece. Right after, a sham therapy was performed, using RAFFAELLO 980 BIO - Dental Medical Technologies - DMT S.r.l. Although the device was switched on, the hand piece did not work and the sound was emitted by a mobile phone. The tip of the laser device was positioned on two areas for each dental element, located one in the center of the cervical region and the other in the middle third of the crown.
  Interventions: Other: CPP-ACPF
- Group B (placebo mousse + PBMT) (Placebo Comparator): A placebo mousse (Elmex Junior®) was applied with a microbrush on the cervical buccal surface of each tooth for 5 minutes and it was subsequently distributed for 20 seconds with a rubber cup coupled to a low speed handpiece. Right after, a PBMT was performed, using RAFFAELLO 980 BIO - Dental Medical Technologies - DMT S.r.l. The tip of the laser device was positioned on two areas for each dental element, located one in the center of the cervical region and the other in the middle third of the crown. The parameters used were: wavelength 980 nm, power 4 W, irradiation area1 cm2, application time 15 sec per 1 cm2, energy density 60 J/cm2
  Interventions: Other: PBMT
- Group C (CPP-ACPF + PBMT) (Experimental): CPP-ACPF mousse (MI Paste®) was applied with a microbrush on the cervical buccal surface of each tooth for 5 minutes and it was subsequently distributed for 20 seconds with a rubber cup coupled to a low speed handpiece. Right after, a PBMT was performed, using RAFFAELLO 980 BIO - Dental Medical Technologies - DMT S.r.l. The tip of the laser device was positioned on two areas for each dental element, located one in the center of the cervical region and the other in the middle third of the crown. The parameters used were: wavelength 980 nm, power 4 W, irradiation area1 cm2, application time 15 sec per 1 cm2, energy density 60 J/cm2
  Interventions: Other: CPP-ACPF+PBMT

INTERVENTIONS:
Other: CPP-ACPF — CPP-ACPF mousse (MI Paste®) was applied with a microbrush on the cervical buccal surface of each tooth for 5 minutes and it was subsequently distributed for 20 seconds with a rubber cup coupled to a low speed handpiece. Right after, a sham therapy was performed, using RAFFAELLO 980 BIO - Dental Medical Technologies - DMT S.r.l. Although the device was switched on, the hand piece did not work and the sound was emitted by a mobile phone. The tip of the laser device was positioned on two areas for each dental element, located one in the center of the cervical region and the other in the middle third of the crown.
  Arms: Group A (CPP-ACPF mousse + sham light therapy)
Other: PBMT — A placebo mousse (Elmex Junior®) was applied with a microbrush on the cervical buccal surface of each tooth for 5 minutes and it was subsequently distributed for 20 seconds with a rubber cup coupled to a low speed handpiece. Right after, a PBMT was performed, using RAFFAELLO 980 BIO - Dental Medical Technologies - DMT S.r.l. The tip of the laser device was positioned on two areas for each dental element, located one in the center of the cervical region and the other in the middle third of the crown. The parameters used were: wavelength 980 nm, power 4 W, irradiation area1 cm2, application time 15 sec per 1 cm2, energy density 60 J/cm2
  Arms: Group B (placebo mousse + PBMT)
Other: CPP-ACPF+PBMT — CPP-ACPF mousse (MI Paste®) was applied with a microbrush on the cervical buccal surface of each tooth for 5 minutes and it was subsequently distributed for 20 seconds with a rubber cup coupled to a low speed handpiece. Right after, a PBMT was performed, using RAFFAELLO 980 BIO - Dental Medical Technologies - DMT S.r.l. The tip of the laser device was positioned on two areas for each dental element, located one in the center of the cervical region and the other in the middle third of the crown. The parameters used were: wavelength 980 nm, power 4 W, irradiation area1 cm2, application time 15 sec per 1 cm2, energy density 60 J/cm2.
  Arms: Group C (CPP-ACPF + PBMT)

SUMMARY:
The aim of this study was to evaluate the efficacy of the association of casein phosphopeptide plus amorphous calcium phosphate (CPP-ACPF) mousse and photo-bio-modulation therapy (PMBT) (diode laser, RAFFAELLO 980 BIO - Dental Medical Technologies - DMT S.r.l.) in the treatment of dental hypersensitivity (DH) in children with Molar Incisor Hypomineralization (MIH) .

Children aged 6-14 years with hypersensitive teeth were randomized into 3 groups. Group A received the application of CPP-ACPF mousse (GC MI Paste®) and sham light therapy; group B got the application of placebo mousse (Elmex Junior®) and PMBT; group C received both CPP-ACPF mousse and PMBT.

DETAILED DESCRIPTION:
Three desensitizing treatment sessions for each group (group A, group B, group C) were performed with a 7 days-interval. The detailed protocol for each treatment is described below.

Group A (CPP-ACPF mousse + sham light therapy) CPP-ACPF mousse (GC MI Paste®) was applied with a microbrush on the cervical buccal surface of each tooth for 5 minutes and it was subsequently distributed for 20 seconds with a rubber cup coupled to a low speed handpiece. Right after, a sham therapy was performed, using RAFFAELLO 980 BIO - Dental Medical Technologies - DMT S.r.l. Although the device was switched on, the hand piece did not work and the sound was emitted by a mobile phone. The tip of the laser device was positioned on two areas for each dental element, located one in the center of the cervical region and the other in the middle third of the crown.

Group B (placebo mousse + PBMT) A placebo mousse (Elmex Junior®) was applied with a microbrush on the cervical buccal surface of each tooth for 5 minutes and it was subsequently distributed for 20 seconds with a rubber cup coupled to a low speed handpiece. Right after, a PBMT was performed, using RAFFAELLO 980 BIO - Dental Medical Technologies - DMT S.r.l. The tip of the laser device was positioned on two areas for each dental element, located one in the center of the cervical region and the other in the middle third of the crown. The parameters used were: wavelength 980 nm, power 4 W, irradiation area1 cm2, application time 15 sec per 1 cm2, energy density 60 J/cm2

Group C (CPP-ACPF + PBMT) CPP-ACPF mousse (GC MI Paste®) was applied with a microbrush on the cervical buccal surface of each tooth for 5 minutes and it was subsequently distributed for 20 seconds with a rubber cup coupled to a low speed handpiece. Right after, a PBMT was performed, using RAFFAELLO 980 BIO - Dental Medical Technologies - DMT S.r.l. The tip of the laser device was positioned on two areas for each dental element, located one in the center of the cervical region and the other in the middle third of the crown. The parameters used were: wavelength 980 nm, power 4 W, irradiation area1 cm2, application time 15 sec per 1 cm2, energy density 60 J/cm2

ELIGIBILITY:
Inclusion Criteria:

* children 6-14 years old
* having at least one MIH-affected tooth and MIH-associated hypersensitivity.

Exclusion Criteria:

* allergy to milk proteins
* chronic diseases,
* carious lesions on the sensitive teeth
* restorations on the sensitive teeth
* other enamel defects (fluorosis, amelogenesis/dentinogenesis imperfecta…)
* presence of orthodontic appliance
* recent anti-inflammatory or cortisone therapies
* recent desensitizing treatments.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-02-10 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Treatment of dental hypersensitivity (DH) | 12 months
  The efficacy of the treatment of dental hypersensitivity was evaluated using the Visual Analogue Scale (VAS), ranging from 0 to 10, with 0=no pain and 10= worst possible pain. The evaluation was performed at the following time points: before (T0) and after (T1) the first session, after the second session (T2) on the 7th day, after the third session (T3) on the 14th day and after 4 weeks from the starting (T4) on the 28th day.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Bardellini, AP, Principal Investigator — Università degli Studi di Brescia
Locations (1):
- Dental Clinic, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No